CLINICAL TRIAL: NCT03378323
Title: Single Versus Multiple Injections for Axillary Plexus Block: a Randomized Controlled Trial
Brief Title: Single Versus Multiple Injections for Axillary Plexus Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hôpital du Valais (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Sina Grape, Dr, Hôpital du Valais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAX Unique
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Upper Extremity
Keywords: upper extremity surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple injection local anesthetic (Active Comparator): Ultrasound guided axillary plexus block with multiple injections of local anesthetic
  Interventions: Drug: Multiple injection local anesthetic
- Single injection local anesthetic (Experimental): Ultrasound guided axillary plexus block with a single injection of local anesthetic
  Interventions: Drug: Single injection local anesthetic

INTERVENTIONS:
Drug: Multiple injection local anesthetic — Multiple injection local anesthetic
  Arms: Multiple injection local anesthetic
Drug: Single injection local anesthetic — Single injection local anesthetic
  Arms: Single injection local anesthetic

SUMMARY:
Patients will be randomized to one of two groups:

1. Multiple injection group: Axillary brachial plexus block with multiple injections, with the arm abducted, performed with the aid of ultrasound;
2. Single injection group: Axillary brachial plexus block with a single injection, with the arm placed behind the head and the elbow flexed, performed with the aid of ultrasound

DETAILED DESCRIPTION:
The study will be proposed to all patients undergoing formarm or hand surgery under axillary brachial plexus block. Patients will be randomized to one of two groups The first group - multiple injection group - will receive an ultrasound-guided axillary brachial plexus block with the traditional technique, i.e. multiple injections of local anesthetic in proximity to the 4 nerfs that innervate the arm. The arm will be abducted during the block procedure.

The second group - single injection group - will receive an ultrasound-guided axillary brachial plexus block with the arm placed behind the head and the elbow flexed. In this position the different nerfs group around the axillary artery where they will be blocked with a single injection of local anesthetic.

All patients will receive the same type and amount of local anesthetic: 30 ml of a mixture of ropivacaine 0.5 % + mepivacaine 1 %.

The primary outcome measure is the time needed for the performance of the block. Secondary outcomes are: success rate of the block at 30 minutes after the injection, needling time, time to first analgesic request, postoperative opioid consumption, pain scores at 12 and 24 hours postoperatively, block-related complications, and patient satisfaction. These outcomes are further defined in the section below.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who undergo forearm or hand surgery under axillary brachial plexus block

Exclusion Criteria:

* History of allergic reaction to local anaesthetics
* Peripheral neuropathy
* Renal or hepatic insufficiency
* Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Performance time | 10 minutes
  Time in minutes from ultrasound probe placement to end of local anesthetic injection

SECONDARY OUTCOMES:
Needling time | 15 minutes
  Time in seconds to complete the block
Time to first analgesic request | 24 hours
  Time in minutes to first analgesic request postoperatively
Block-related complications | 24 hours
  Infection, bleeding, neurological problems, pain during the 24 postoperative hours
Postoperative opioid consumption on postoperative day 1 | 24 hours
  intravenous morphine equivalent consumption during the 24 postoperative hours
Pain scores at 12 hours postoperatively | 12 hours
  Measured on a visual analogue scale between 0 and 10 (0 = no pain, 10 = worst pain imaginable)
Pain scores on postoperative day 1 | 24 hours
  Measured on a visual analogue scale between 0 and 10 (0 = no pain, 10 = worst pain imaginable)
Patient satisfaction | 24 hours
  Assessed by numerical rating scale on a scale between 0 (= completely dissatisfied) and 10 (= completely satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Sina Grape, MD, Principal Investigator — Hôpital du Valais; Eric Albrecht, MD, Study Director — University of Lausanne Hospitals
Locations (1):
- Hopital du Valais, Sion, Switzerland